CLINICAL TRIAL: NCT03157674
Title: Real-World Evidence and Treatment Patterns: Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-868
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Head & Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- HNC patients: HNC patients who have been diagnosed with HNC between
  01-Jan-2013 and 30-Sep-2016.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study will be focused on HNC patients who have been diagnosed with HNC between 01-Jan-2013 and 30-Sep-2016.

ELIGIBILITY:
Inclusion Criteria:

* HNC or undefined histology (not otherwise specified [NOS]) HNC diagnosis from 01-Jan-2013 to 30-Sep-2016 using Japanese disease code
* Age 18 years or older at initial diagnosis of HNC regardless of staging

Exclusion Criteria:

* Diagnosis of another malignancy on or before the initial diagnosis of HNC with the exception of non-melanoma skin cancer and metastatic cancer
* Diagnosis of HNC before 01-Jan 2013 or after 30-Sep-2016

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Medical Data Vision (MDV) database with a HNC diagnosis will be used to identify eligible subjects by applying the patient inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 43994 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving radiotherapy as anti-cancer treatment | Approximately 45 months
Proportion of patients receiving surgery as anti-cancer treatment | Approximately 45 months
Proportion of patients receiving chemotherapy as anti-cancer treatment | Approximately 45 months
Proportion of patients receiving targeted therapy as anti-cancer treatment | Approximately 45 months
Proportion of patients receiving supportive care as anti-cancer treatment | Approximately 45 months
Distribution of Treatment History in Head and Neck Cancer (HNC) patients | Approximately 45 months

SECONDARY OUTCOMES:
Distribution of overall survival (OS) by age | Approximately 45 months
Distribution of overall survival (OS) by gender | Approximately 45 months
Distribution of overall survival (OS) by stage | Approximately 45 months
Distribution of overall survival (OS) by tumor site | Approximately 45 months
Distribution of overall survival (OS) by treatment regimen | Approximately 45 months
Number of treatment-limiting adverse events (AEs) | Approximately 45 months
  Incidence of important treatment-limiting adverse events (AEs) associated with systemic therapies
Number of withdrawals due to AEs | Approximately 45 months
Proportion of diagnosis of another malignancy on or before the initial diagnosis of HNC | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tokyo, Shibuya-ku, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm